CLINICAL TRIAL: NCT03607617
Title: ASCEND: ApproacheS to CHC ImplEmeNtation of SDH Data Collection and Action
Acronym: ASCEND
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: OCHIN, Inc. (Other); Oregon Health and Science University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1R18DK114701-01 (NIH); 1R18DK114701-01 (NIH)
Record Dates: First submitted 2018-06-01; First posted 2018-07-31 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus
Keywords: social determinants of health; community health clinic; primary care; electronic medical record
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Wedge 1: 4 randomized clinics will implement SDH tool.
  Interventions: Other: SDH Tool
- Wedge 2: 5 randomized clinics implement SDH tool 24 weeks following prior wedge implementation.
  Interventions: Other: SDH Tool
- Wedge 3: 5 randomized clinics implement SDH tool 24 weeks following prior wedge implementation.
  Interventions: Other: SDH Tool
- Wedge 4: 5 randomized clinics implement SDH tool 24 weeks following prior wedge implementation.
  Interventions: Other: SDH Tool
- Wedge 5: 6 randomized clinics implement SDH tool 24 weeks following prior wedge implementation.
  Interventions: Other: SDH Tool
- Wedge 6: 6 randomized clinics implement SDH tool 24 weeks following prior wedge implementation.
  Interventions: Other: SDH Tool

INTERVENTIONS:
Other: SDH Tool — The SDH tool is embedded in the EMR to collect and act on individualized social determinants of health data.

SUMMARY:
This work will test a set of strategies for helping community health centers (CHCs) routinely identify and take action on the SDH-related needs of patients with / at risk for DM using a stakeholder-driven process to develop EHR-based SDH data collection / summary tools for CHCs.

DETAILED DESCRIPTION:
This work will test a set of strategies for helping community health centers(CHCs) routinely identify and take action on the SDH-related needs of patients with / at risk for DM. The work will specifically study: (a) EHR-based SDH data collection / action in CHCs, and (b) the impact of a set of scalable implementation strategies known to support clinical practice changes (the 'SDH Action Plan'), on CHCs' adoption of SDH data collection and action. Focusing on DM risk management and obesity prevention outcomes in adult patients, the investigators will conduct a mixed methods formative evaluation of SDH data collection uptake among CHCs that had SDH data tools activated in their EHR in June 2016. (Quantitative data will come from all 440 CHCs' shared EHR, qualitative data from 10-12 CHCs purposively recruited from this pool). Identify patterns of SDH data collection in these diverse CHCs, and clinic-level factors associated with variation in SDH data collection rates. Use results to fine-tune the SDH Action Plan intervention's strategies for helping CHCs systematically: (i) collect SDH data in standard workflows, and (ii) integrate SDH data into care plans (e.g., making referrals to social services; adapting treatment plans) for adults with / at risk for DM.

Through a pragmatic, stepped-wedge, cluster-randomized trial in 30 CHCs, the CHCs will be randomized to one of five 6-month wedges, with staggered timing. CHCs in each wedge will receive intensive implementation support (the SDH Action Plan). This scalable intervention includes both comprehensive technical assistance and training materials designed to help CHCs plan for and implement SDH data collection / action, and six months of remote access to an 'SDH Implementation Team' that will tailor implementation support to each CHC's needs, with an emphasis on the Building Blocks of Primary Care.45 To test this approach, the investigators will conduct a realist evaluation of whether and how the SDH Action Plan intervention improves: (i) SDH data collection in CHC workflows; (ii) integration of SDH data into DM risk management care; and (iii) clinical measures associated with effective DM risk management (controlled blood pressure, HbA1c, BMI, lipids, etc.; up-to-date preventive care). H3a: Intervention CHCs will have significantly greater increases in (i) SDH data collection, and (ii) actions taken to address SDH needs, compared to control CHCs. H3b: Patients at intervention CHCs for whom SDH data are collected will have significant improvements in DM / obesity risk management / receipt of related preventive care, compared to those at control CHCs.

ELIGIBILITY:
Inclusion Criteria:

* Any persons who are at risk for type 2 diabetes
* May include some subjects with mental health conditions of various types; however, it is important to systematically address high DM /obesity risk in this population, because such patients may be at risk for elevated high DM /obesity risk and have often been excluded or underrepresented in previous research studies.
* Decisionally/cognitively impaired
* Economically/educationally disadvantaged
* Non-English Speakers
* Elderly

Exclusion Criteria:

* Neonates of uncertain viability or nonviable neonates (up to 28 days post birth)
* Prisoners

Note: The investigators are not enrolling patients for this clinic-randomized study, but rather studying the uptake and impact of a set of EHR-based clinical decision support tools into regular care at the participating clinics. In this clinic-randomized trial, the intervention / randomization are clinic level. The intervention targets clinic processes that are part of the regular care patients receive, and will not require special visits.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any persons who are at risk for type 2 diabetes seen at the participating study CHC.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Gold, PhD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gold R, Kaufmann J, Gottlieb LM, Weiner SJ, Hoopes M, Gemelas JC, Torres CH, Cottrell EK, Hessler D, Marino M, Sheppler CR, Berkowitz SA. Cross-Sectional Associations: Social Risks and Diabetes Care Quality, Outcomes. Am J Prev Med. 2022 Sep;63(3):392-402. doi: 10.1016/j.amepre.2022.03.011. Epub 2022 May 4. PMID 35523696
- [Derived] Haley AD, Powell BJ, Walsh-Bailey C, Krancari M, Gruss I, Shea CM, Bunce A, Marino M, Frerichs L, Lich KH, Gold R. Strengthening methods for tracking adaptations and modifications to implementation strategies. BMC Med Res Methodol. 2021 Jun 26;21(1):133. doi: 10.1186/s12874-021-01326-6. PMID 34174834
- [Derived] Gold R, Bunce A, Cottrell E, Marino M, Middendorf M, Cowburn S, Wright D, Mossman N, Dambrun K, Powell BJ, Gruss I, Gottlieb L, Dearing M, Scott J, Yosuf N, Krancari M. Study protocol: a pragmatic, stepped-wedge trial of tailored support for implementing social determinants of health documentation/action in community health centers, with realist evaluation. Implement Sci. 2019 Jan 28;14(1):9. doi: 10.1186/s13012-019-0855-9. PMID 30691480

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol enrollment (n=31) describes the number of clinics enrolled in the study. Number of participants describes the patients of participating clinics used for analysis. The total number of patients in the completed row after duplicate records are removed is 358,818.
Units Other Than Participants: Number of Clinics
Groups:
- Wedge 1: 1) 6 months pre-intervention, 2) 6 months SDH intervention, 3) 36 months post-intervention monitoring
- Wedge 2: 1) 12 months pre-intervention, 2) 6 months SDH intervention, 3) 30 months post-intervention monitoring
- Wedge 3: 1) 18 months pre-intervention, 2) 6 months SDH intervention, 3) 24 months post-intervention monitoring
- Wedge 4: 1) 24 months pre-intervention, 2) 6 months SDH intervention, 3) 18 months post-intervention monitoring
- Wedge 5: 1) 30 months pre-intervention, 2) 6 months SDH intervention, 3) 12 months post-intervention monitoring
- Wedge 6: 1) 36 months pre-intervention, 2) 6 months SDH intervention, 3) 6 months post-intervention monitoring
Period: Overall Study
Arm/Group | Wedge 1 | Wedge 2 | Wedge 3 | Wedge 4 | Wedge 5 | Wedge 6
Started | 24650; 4 Number of Clinics | 108752; 5 Number of Clinics | 21743; 5 Number of Clinics | 66504; 5 Number of Clinics | 64082; 6 Number of Clinics | 122138; 6 Number of Clinics
Step 1: 1-6 Months (Wedge 1 Intervention Started 9/2018) | 24650; 4 Number of Clinics | 0; 0 Number of Clinics | 0; 0 Number of Clinics | 0; 0 Number of Clinics | 0; 0 Number of Clinics | 0; 0 Number of Clinics
Step 2: 7-12 Months (Wedge 2 Intervention Started 3/2019) | 24650; 4 Number of Clinics | 108752; 5 Number of Clinics | 0; 0 Number of Clinics | 0; 0 Number of Clinics | 0; 0 Number of Clinics | 0; 0 Number of Clinics
Step 3: 13-18 Months (Wedge 3 Intervention Started 9/2019) | 24650; 4 Number of Clinics | 108752; 5 Number of Clinics | 21743; 5 Number of Clinics | 0; 0 Number of Clinics | 0; 0 Number of Clinics | 0; 0 Number of Clinics
Step 4: 19-24 Months (Wedge 4 Intervention Started 2/2020) | 24650; 4 Number of Clinics | 108752; 5 Number of Clinics | 21743; 5 Number of Clinics | 66504; 5 Number of Clinics | 0; 0 Number of Clinics | 0; 0 Number of Clinics
Step 5: 25-30 Months (Wedge 5 Intervention Started 8/2020) | 24650; 4 Number of Clinics | 108752; 5 Number of Clinics | 21743; 5 Number of Clinics | 66504; 5 Number of Clinics | 64082; 6 Number of Clinics | 0; 0 Number of Clinics
Step 6: 31-36 Months (Wedge 6 Intervention Started 1/2021) | 24650; 4 Number of Clinics | 108752; 5 Number of Clinics | 21743; 5 Number of Clinics | 66504; 5 Number of Clinics | 64082; 6 Number of Clinics | 122138; 6 Number of Clinics
Completed | 24650; 4 Number of Clinics | 108752; 5 Number of Clinics | 21743; 5 Number of Clinics | 66504; 5 Number of Clinics | 64082; 6 Number of Clinics | 122138; 6 Number of Clinics
Not Completed | 0; 0 Number of Clinics | 0; 0 Number of Clinics | 0; 0 Number of Clinics | 0; 0 Number of Clinics | 0; 0 Number of Clinics | 0; 0 Number of Clinics

BASELINE CHARACTERISTICS:
Population: Number of patients at the participating clinics for each wedge. If a patient was in more than one wedge (many patients had visits at different clinics), the patient will be counted more than once in the "Total" column. Note: the "Baseline Analysis Population" Total column is a calculated field that cannot be revised. 358,818 patients were analyzed (after duplicates removed).
Units Other Than Participants: Clinics
Groups:
- Total: Total of all reporting groups
Arm/Group | Wedge 1 | Wedge 2 | Wedge 3 | Wedge 4 | Wedge 5 | Wedge 6 | Total
Number analyzed (Participants) | 24650 | 108752 | 21743 | 66504 | 64082 | 122138 | 407869
Number analyzed (Clinics) | 4 | 5 | 5 | 5 | 6 | 6 | 31
Age, Continuous [Median (Full Range); unit: years] — Age by Wedge. If a patient was in more than one wedge (many patients had visits at different clinics), the patient will be counted more than once in the "Total analyzed" column.
  years | 36 [24 to 47] | 44 [43 to 50] | 45 [29 to 46] | 45 [39 to 55] | 44 [35 to 53] | 45 [41 to 57] | 45 [24 to 57]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex/Gender by Wedge. If a patient was in more than one wedge (many patients had visits at different clinics), the patient will be counted more than once in the "Total analyzed" column.
  Participants
    Female | 11787 | 60088 | 11299 | 36452 | 32026 | 67403 | 219055
    Male | 12839 | 48627 | 10436 | 30011 | 32017 | 54675 | 188605
    Unknown | 24 | 37 | 8 | 41 | 39 | 60 | 209
Race/Ethnicity, Customized [Number; unit: Percent] — Race/Ethnicity by Wedge. If a patient was in more than one wedge (many patients had visits at different clinics), the patient will be counted more than once in the "Total" column.
  Percent
    Hispanic | 10 | 35.3 | 24.5 | 26.8 | 17.4 | 44.8 | 33
    Non-Hispanic Black | 61.3 | 6.6 | 43 | 7.1 | 20.7 | 6 | 13.1
    Non-Hispanic, non-Black, nonwhite | 9.6 | 7.3 | 3.2 | 3.8 | 3.8 | 4.2 | 5
    Non-Hispanic white | 17.5 | 43.9 | 22.9 | 49.4 | 49.4 | 35.9 | 40.5
    Not documented in EHR | 1.6 | 7 | 6.4 | 12.9 | 8.6 | 9 | 8.3

OUTCOME MEASURES:

1. Primary Outcome: Social Risk Screening
Description: Average differences are reported comparing the pre-intervention period (6 months or more) to (1) the six-month intervention period and (2) the post-intervention period (6 months or more). Numerator is measured as the number of patients with documented social risk screening results entered at a clinical encounter in the measurement period (excluding those only for COVID-19 testing/vaccination, as many people received these services at the study sites who were not otherwise patients at these clinics). Denominator is total patients seen in that period. Domains of social risk screening included child/family care insecurity, education, employment, financial strain, food insecurity, health insurance, health literacy, housing instability, inadequate physical activity, relationship safety, social isolation, stress, transportation needs, and utilities insecurity.
Time Frame: During 6-month intervention and postintervention (6 months or more, all months from the intervention period's end through December 2021)
Measure: Number (95% Confidence Interval); unit: Rate Ratio (RR)
Groups:
- During 6-month Intervention; Postintervention: Added effects of intervention compared with preintervention, RR (95% CI)
Arm/Group | During 6-month Intervention | Postintervention
Number analyzed (Participants) | 155747 | 241606
Rate Ratio (RR) | 2.45 [1.32 to 4.39] | 2.16 [0.64 to 7.27]

2. Secondary Outcome: Social Risk Referral
Description: Average differences are reported comparing the pre-intervention period (6 months or more) to (1) the six-month intervention period and (2) the post-intervention period (6 months or more). Monthly clinic rate of provision of social risk-related referrals, measured as the number of patients with a documented referral among all patients seen in the measurement period (regardless of whether social risk screening was documented). This outcome included referrals internal (e.g., to a social worker) or external (e.g., to housing services) to the clinic. Denominator is total patients seen in that period.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Rate Ratio (RR)
Arm/Group | During 6-month Intervention | Postintervention
Number analyzed (Participants) | 155747 | 241606
Rate Ratio (RR) | 1.33 [0.73 to 2.43] | 0.89 [0.18 to 1.93]

3. Secondary Outcome: Control of DM Risk Management Biomarkers: Blood Pressure (BP)
Description: Average differences are reported comparing the pre-intervention period (6 months or more) to (1) the six-month intervention period and (2) the post-intervention period (6 months or more). Numerator is measured as the percent of patients with BP controlled (<140/80 mmHg)--measured with systolic and diastolic pressure, denominator is total patients seen in that period with the needed follow-up data. This table is a subpopulation cohort comprised of patients with an encounter during the study period and established diabetes before the second month of their clinic's baseline period (excluding pregnant women).
Time Frame: as for outcome 1
Population: This table is a subpopulation cohort comprised of patients with an encounter during the study period and established diabetes before the second month of their clinic's baseline period (excluding pregnant women).
Measure: Number (95% Confidence Interval); unit: Percent controlled
Groups:
- During 6-month Intervention; Postintervention: Added effects associated with intervention compared with preintervention, absolute percent change (95% CI)
Arm/Group | During 6-month Intervention | Postintervention
Number analyzed (Participants) | 155747 | 241606
Percent controlled
  Patients with diabetes screened for social risks (subset): number analyzed (Participants) | 15783 | 23190
  Patients with diabetes screened for social risks (subset) | 1.35 [-1.96 to 4.65] | 11.26 [1.51 to 21.00]
  All patients with diabetes | -0.90 [-3.37 to 1.56] | 1.57 [-6.21 to 9.36]

4. Secondary Outcome: Control of DM Risk Management Biomarkers: HbA1c
Description: Average differences are reported comparing the pre-intervention period (6 months or more) to (1) the six-month intervention period and (2) the post-intervention period (6 months or more). Numerator is measured as the percent of patients with A1c controlled (<7.0%), denominator is total patients seen in that period with the needed follow-up data. This table is a subpopulation cohort comprised of patients with an encounter during the study period and established diabetes before the second month of their clinic's baseline period (excluding pregnant women).
Time Frame: During 6-month intervention and postintervention (6-months or more, all months from the intervention period's end through December 2021)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percent controlled
Arm/Group | During 6-month Intervention | Postintervention
Number analyzed (Participants) | 155747 | 241606
Percent controlled
  Patients with diabetes screened for social risks (subset): number analyzed (Participants) | 10431 | 20642
  Patients with diabetes screened for social risks (subset) | -2.01 [-7.50 to 3.47] | -6.74 [-15.98 to 2.49]
  All patients with diabetes | -2.05 [-5.26 to 1.17] | -6.46 [-13.52 to 0.61]

5. Secondary Outcome: Control of DM Risk Management Biomarkers: LDL
Description: Average differences are reported comparing the pre-intervention period (6 months or more) to (1) the six-month intervention period and (2) the post-intervention period (6 months or more). Numerator is measured as the percent of patients with Low-density lipoprotein (LDL) controlled (l<100 mg/dL), denominator is total patients seen in that period with the needed follow-up data. This table is a subpopulation cohort comprised of patients with an encounter during the study period and established diabetes before the second month of their clinic's baseline period (excluding pregnant women).
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percent controlled
Arm/Group | During 6-month Intervention | Postintervention
Number analyzed (Participants) | 155747 | 241606
Percent controlled
  Patients with diabetes screened for social risks (subset): number analyzed (Participants) | 4672 | 17824
  Patients with diabetes screened for social risks (subset) | 4.19 [-1.86 to 10.25] | 7.33 [-2.61 to 17.27]
  All patients with diabetes | 4.63 [-0.05 to 9.30] | 5.61 [-2.99 to 14.20]

6. Secondary Outcome: DM Key Tests (Screening, Percent up to Date)
Description: Average differences are reported comparing the pre-intervention period (6 months or more) to (1) the six-month intervention period and (2) the post-intervention period (6 months or more). Numerator is measured as the rate of patients with up-to-date on DM key tests (annual low-density lipoprotein (LDL), biannual hemoglobin A1C (HbA1c)), denominator is total patients seen in that period with the needed follow-up data. This table is a subpopulation cohort comprised of patients with an encounter during the study period and established diabetes before the second month of their clinic's baseline period (excluding pregnant women).
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: screen, % up to date
Arm/Group | During 6-month Intervention | Postintervention
Number analyzed (Participants) | 155747 | 241606
screen, % up to date
  HbA1c (patients with diabetes screened for social risks (subset)): number analyzed (Participants) | 26252 | 26252
  HbA1c (patients with diabetes screened for social risks (subset)) | -7.50 [-14.51 to -0.49] | -23.26 [-48.13 to 1.62]
  HbA1c (all patients with diabetes) | -9.92 [-15.91 to -3.94] | -30.51 [-50.20 to -10.83]
  LDL (patients with diabetes screened for social risks (subset)): number analyzed (Participants) | 26252 | 26252
  LDL (patients with diabetes screened for social risks (subset)) | -8.53 [-15.03 to -2.02] | -29.95 [-54.58 to -5.32]
  LDL (all patients with diabetes) | -10.02 [-15.75 to -4.30] | -33.20 [-54.01 to -12.39]

ADVERSE EVENTS:
Description: Adverse events were not monitored or assessed. ASCEND is a minimal risk study because it tests whether an implementation support intervention (6 months of technical assistance and coaching) to clinics improves the adoption of social risk activities as part of standards of care. Therefore, there were no adverse risks to patients involved in this study beyond data management risks (e.g. breach of confidentiality).
Arm/Group | Wedge 1 | Wedge 2 | Wedge 3 | Wedge 4 | Wedge 5 | Wedge 6
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT03607617/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT03607617/SAP_001.pdf